CLINICAL TRIAL: NCT02522728
Title: Evaluation of Triathlon - A New Total Knee Prosthesis System - Roentgen Stereophotogrammetric Analysis Triathlon CR vs. PS
Brief Title: Evaluation of Triathlon - A New Total Knee Prosthesis System - Roentgen Stereophotogrammetric Analysis (RSA) Triathlon CR vs. PS
Acronym: TriathlonRSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K-S-015 Triathlon RSA _2
Record Dates: First submitted 2015-06-11; First posted 2015-08-13 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Knee; Arthroplasty; Implant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triathlon CR (Active Comparator): Triathlon Cruciate Retaining (CR) versus Triathlon Posterior Stabilized (PS): During knee prosthesis surgery the surgeon many times need to make a judgement on if to keep a defect anatomical structure or if to replace it with knee prosthesis with a design that allows for adjustment of this defect. This study is aimed to evaluate which prosthetic choice to be made in respect of stability, long-term results and patient outcome.
  Interventions: Device: Triathlon CR
- Triathlon PS (Active Comparator): Triathlon Cruciate Retaining (CR) versus Triathlon Posterior Stabilized (PS): During knee prosthesis surgery the surgeon many times need to make a judgement on if to keep a defect anatomical structure or if to replace it with knee prosthesis with a design that allows for adjustment of this defect. This study is aimed to evaluate which prosthetic choice to be made in respect of stability, long-term results and patient outcome.
  Interventions: Device: Triathlon PS

INTERVENTIONS:
Device: Triathlon CR — Implantation of Knee Prosthesis
  Arms: Triathlon CR
Device: Triathlon PS — Implantation of Knee Prosthesis
  Arms: Triathlon PS

SUMMARY:
The objective is to investigate the Clinical, Radiographic, Roentgen Stereophotogrammetric behaviour and patient outcome when using the Triathlon total knee prosthesis in a prospective randomized clinical trial.

DETAILED DESCRIPTION:
The objective is to investigate the Clinical, Radiographic, Roentgen Stereophotogrammetric behaviour and patient outcome when using the Triathlon total knee prosthesis in a prospective randomized clinical trial.

The evaluation is carried out by a prospective randomised RSA-study with Triathlon CR vs. Triathlon PS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffering exclusively from osteo arthritis, Stage II-V [Ahlbäck, 1968 391] will be operated.
2. Patients requiring knee prosthesis, suitable for the use of Duracon and Triathlon knee system
3. Patients who understand the conditions of the study and are willing and able to comply with the post-operative scheduled clinical and radiographical evaluations and the prescribed rehabilitation.
4. Patients who signed the Ethics Committee approved Informed Consent Form prior to surgery.

Exclusion Criteria:

1. Previous major knee surgery
2. Other significant disabling problems from the muscular-skeletal system than in the knees
3. Obese patients where obesity is severe enough to affect subject's ability to perform activities of daily living (body mass index, kg/m2: BMI above 35).
4. Patients with active or suspected infection.
5. Patients with malignancy - active malignancy.
6. Patients with severe osteoporosis, Paget's disease, renal osteodystrophy.
7. Patients immunologically suppressed, or receiving steroids in excess of physiologic dose requirements.
8. The patient has a neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device or the patient has a neurological deficit which interferes with the patient's ability to limit weight bearing or places an extreme load on the implant during the healing period.
9. Female patients planning a pregnancy during the course of the study.
10. Patients with systemic or metabolic disorders leading to progressive bone deterioration.
11. Patients, who as judged by the surgeon, are mentally incompetent or are unlikely to be compliant with the prescribed post-operative routine and follow-up evaluation schedule.
12. Patients with other severe concurrent joint involvements, which can affect their outcome.
13. Patients with other concurrent illnesses, which are likely to affect their outcome such as sickle cell anaemia, systemic lupus erythematosus or renal disease requiring dialysis.
14. Patients under the protection of law (e.g. guardianship).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-01-23 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sören Toksvig-Larsen, MD, Principal Investigator — Skånevård Kryh Division Kirurgi och Ortopedkliniken Hässleholm
Locations (1):
- Skånevård Kryh Division Kirurgi och Ortopedkliniken Hässleholm, Hässleholm, Skåne County, Sweden

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Triathlon CR | Triathlon PS
Started | 28 | 30
Completed | 16 | 19
Not Completed | 12 | 11
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Death | 4 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Did not receive randomized study device | 0 | 1

BASELINE CHARACTERISTICS:
Population: With an alpha of 0.05 and a beta of 0.20 the required sample size in each group is 25 patients. Patients with inadequate marking will be excluded from the study. Taking the latter into account and to compensate for possible lost to follow up, 30 patients will be recruited per study group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Triathlon CR | Triathlon PS | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.07 (8.11) | 67.47 (7.64) | 67.77 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 9 | 14 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 28 | 30 | 58
Ahlbäck Classification [Count of Participants; unit: Participants] — According to Ahlbäck system, knee joint osteoarthritis is classified as:
  grade 1: joint space narrowing (less than 3 mm) grade 2: joint space obliteration grade 3: minor bone attrition (0-5 mm) grade 4: moderate bone attrition (5-10 mm) grade 5: severe bone attrition (more than 10 mm)
  Participants
    Grade 1 | 0 | 0 | 0
    Grade 2 | 8 | 18 | 26
    Grade 3 | 20 | 12 | 32
    Grade 4 | 0 | 0 | 0
    Grade 5 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Fixation and Stability of the Triathlon Total Knee Prosthesis by Roentgen Stereophotogrammetric Analysis (RSA)
Description: Roentgen Stereophotogrammetric Analysis (RSA) is a technique to measure migration of prosthesis components relative to the bone which allows conclusions regarding the fixation of an implant. This study assesses the fixation and stability of the Triathlon total knee prosthesis at 2 years by RSA as a predictor of late mechanical loosening.
Time Frame: 2 years follow-up
Population: The number included in the analysis differs from the overall number analysed because that data were not collected.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Triathlon CR | Triathlon PS
Number analyzed (Participants) | 22 | 27
mm | 0.68 (0.41) | 0.79 (0.53)

2. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Knee Society Score (KSS)
Description: The Knee Society Clinical Rating System is comprised of two distinct sub-scores: 1. assessment score for pain, range of motion (ROM) and joint stability, 2. score for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Time Frame: pre-operative, 3 months, 1, 2, 5, 7 and 10 years
Population: The number included in the analysis in one or more rows differs from the overall number analysed because that data were not collected.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triathlon CR | Triathlon PS
Number analyzed (Participants) | 28 | 30
units on a scale
  pre-op assessment score | 20.43 (8.37) | 25.5 (7.41)
  3 months assessment score: number analyzed (Participants) | 25 | 30
  3 months assessment score | 91.88 (9.94) | 91.57 (12.65)
  1 year assessment score: number analyzed (Participants) | 24 | 30
  1 year assessment score | 95.00 (7.61) | 94.70 (8.32)
  2 years assessment score: number analyzed (Participants) | 22 | 28
  2 years assessment score | 97.00 (5.41) | 97.39 (4.60)
  5 years assessment score: number analyzed (Participants) | 19 | 24
  5 years assessment score | 95.47 (9.64) | 98.33 (3.42)
  7 years assessment score: number analyzed (Participants) | 17 | 20
  7 years assessment score | 94.12 (11.88) | 98.10 (4.58)
  10 years assessment score: number analyzed (Participants) | 16 | 18
  10 years assessment score | 95.06 (12.57) | 97.78 (6.99)
  pre-op function score | 49.11 (11.71) | 50.67 (12.71)
  3 months function score: number analyzed (Participants) | 25 | 30
  3 months function score | 79.80 (15.10) | 72.17 (17.78)
  1 year function score: number analyzed (Participants) | 24 | 30
  1 year function score | 88.54 (17.41) | 85.00 (16.76)
  2 years function score: number analyzed (Participants) | 22 | 28
  2 years function score | 94.32 (8.49) | 89.46 (15.89)
  5 years function score: number analyzed (Participants) | 19 | 24
  5 years function score | 87.89 (17.27) | 89.79 (17.84)
  7 years function score: number analyzed (Participants) | 17 | 20
  7 years function score | 89.41 (15.70) | 88.00 (16.42)
  10 years function score: number analyzed (Participants) | 16 | 18
  10 years function score | 93.43 (13.26) | 91.39 (13.48)

3. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Knee Injury and Osteoarthritis Outcome Score (KOOS) Patient Questionnaire
Description: KOOS consists of 5 subscales: Pain, other symptoms, function in daily living , function in sport and recreation and knee related quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no problems or a better outcome and 0 indicating extreme problems or a worse outcome).
Time Frame: pre-operative, 3 months, 1, 2, 5, 7 and 10 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triathlon CR | Triathlon PS
Number analyzed (Participants) | 28 | 30
units on a scale
  pre-op symptom: number analyzed (Participants) | 27 | 29
  pre-op symptom | 47.37 (18.19) | 54.66 (20.05)
  3 months symptom: number analyzed (Participants) | 25 | 30
  3 months symptom | 65.67 (17.13) | 66.11 (14.47)
  1 year symptom: number analyzed (Participants) | 23 | 28
  1 year symptom | 75.96 (18.72) | 76.19 (14.99)
  2 years symptom: number analyzed (Participants) | 22 | 28
  2 years symptom | 91.49 (18.46) | 82.78 (15.49)
  5 years symptom: number analyzed (Participants) | 19 | 24
  5 years symptom | 86.47 (19.94) | 87.80 (12.19)
  7 years symptom: number analyzed (Participants) | 17 | 20
  7 years symptom | 82.98 (18.58) | 87.86 (11.73)
  10 years symptom: number analyzed (Participants) | 15 | 20
  10 years symptom | 84.29 (18.30) | 84.82 (14.42)
  pre-op pain: number analyzed (Participants) | 27 | 29
  pre-op pain | 38.79 (18.56) | 43.80 (18.57)
  3 months pain: number analyzed (Participants) | 25 | 30
  3 months pain | 70.11 (15.51) | 71.62 (20.20)
  1 year pain: number analyzed (Participants) | 23 | 28
  1 year pain | 83.77 (14.17) | 79.81 (18.92)
  2 years pain: number analyzed (Participants) | 22 | 28
  2 years pain | 88.01 (17.32) | 87.98 (13.75)
  5 years pain: number analyzed (Participants) | 19 | 24
  5 years pain | 85.53 (23.86) | 90.74 (13.84)
  7 years pain: number analyzed (Participants) | 17 | 20
  7 years pain | 86.37 (24.03) | 88.19 (15.61)
  10 years pain: number analyzed (Participants) | 15 | 20
  10 years pain | 90.88 (17.16) | 88.49 (14.47)
  pre-op ADL: number analyzed (Participants) | 27 | 29
  pre-op ADL | 44.16 (16.16) | 45.07 (14.86)
  3 months ADL: number analyzed (Participants) | 25 | 30
  3 months ADL | 72.28 (14.82) | 73.68 (18.70)
  1 year ADL: number analyzed (Participants) | 23 | 28
  1 year ADL | 83.64 (17.07) | 78.73 (19.86)
  2 years ADL: number analyzed (Participants) | 22 | 28
  2 years ADL | 86.61 (14.21) | 83.85 (15.62)
  5 years ADL: number analyzed (Participants) | 19 | 24
  5 years ADL | 84.06 (20.82) | 87.32 (16.98)
  7 years ADL: number analyzed (Participants) | 17 | 20
  7 years ADL | 84.26 (20.08) | 84.20 (19.31)
  10 years ADL: number analyzed (Participants) | 15 | 20
  10 years ADL | 88.53 (18.61) | 82.82 (18.05)
  pre-op Sport Rec: number analyzed (Participants) | 27 | 29
  pre-op Sport Rec | 18.15 (25.39) | 11.72 (12.77)
  3 months Sport Rec: number analyzed (Participants) | 25 | 28
  3 months Sport Rec | 27.80 (19.16) | 30.70 (24.00)
  1 year Sport Rec: number analyzed (Participants) | 23 | 28
  1 year Sport Rec | 38.91 (21.84) | 37.81 (23.65)
  2 years Sport Rec: number analyzed (Participants) | 22 | 28
  2 years Sport Rec | 41.88 (27.45) | 45.53 (22.21)
  5 years Sport Rec: number analyzed (Participants) | 19 | 24
  5 years Sport Rec | 41.32 (31.26) | 56.46 (29.40)
  7 years Sport Rec: number analyzed (Participants) | 17 | 20
  7 years Sport Rec | 45.88 (30.68) | 44.00 (24.58)
  10 years Sport Rec: number analyzed (Participants) | 15 | 18
  10 years Sport Rec | 52.67 (27.77) | 43.75 (28.37)
  Pre-op QOL: number analyzed (Participants) | 27 | 29
  Pre-op QOL | 21.76 (11.55) | 24.57 (14.46)
  3 months QOL: number analyzed (Participants) | 25 | 28
  3 months QOL | 52.25 (17.29) | 56.47 (22.72)
  1 year QOL: number analyzed (Participants) | 25 | 28
  1 year QOL | 68.84 (18.05) | 67.63 (24.59)
  2 years QOL: number analyzed (Participants) | 22 | 28
  2 years QOL | 77.84 (22.14) | 79.02 (19.70)
  5 years QOL: number analyzed (Participants) | 19 | 24
  5 years QOL | 80.59 (24.99) | 82.55 (18.97)
  7 years QOL: number analyzed (Participants) | 17 | 20
  7 years QOL | 75.54 (25.66) | 81.25 (17.33)
  10 years QOL: number analyzed (Participants) | 14 | 20
  10 years QOL | 64.43 (18.79) | 63.75 (11.93)

4. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With EuroQuol-5 Dimension (EQ-5D) Patient Questionnaire
Description: The EQ-5D is a subject-completed questionnaire designed to assess subject health state values. The EQ-5D consists of 2 areas; EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D descriptive system comprises the following five dimensions: mobility self care, usual activities, pain/comfort and anxiety/depression. Each dimension has 3 levels indicating no problems, some problems or extreme problems. The index values on a scale between -1 (low) and 1 (high) are showing the average health status according to the 5 dimensions: A low score shows worse health and a high score shows better health.
  With the EQ VAS the respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Time Frame: 1, 2, 5, 7 and 10 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triathlon CR | Triathlon PS
Number analyzed (Participants) | 28 | 30
units on a scale
  Descriptive EQ-5D 1 year: number analyzed (Participants) | 21 | 26
  Descriptive EQ-5D 1 year | 0.88 (0.15) | 0.80 (0.12)
  Descriptive EQ-5D 2 years: number analyzed (Participants) | 21 | 27
  Descriptive EQ-5D 2 years | 0.88 (0.15) | 0.89 (0.12)
  Descriptive EQ-5D 5 years: number analyzed (Participants) | 19 | 24
  Descriptive EQ-5D 5 years | 0.85 (0.28) | 0.87 (0.15)
  Descriptive EQ-5D 7 years: number analyzed (Participants) | 17 | 20
  Descriptive EQ-5D 7 years | 0.82 (0.16) | 0.75 (0.35)
  Descriptive EQ-5D 10 years: number analyzed (Participants) | 14 | 20
  Descriptive EQ-5D 10 years | 0.91 (0.16) | 0.90 (0.14)
  EQ-5D VAS 1 year: number analyzed (Participants) | 22 | 27
  EQ-5D VAS 1 year | 84 (14) | 83 (13)
  EQ-5D VAS 2 year: number analyzed (Participants) | 21 | 28
  EQ-5D VAS 2 year | 82 (18) | 84 (16)
  EQ-5D VAS 5 year: number analyzed (Participants) | 19 | 24
  EQ-5D VAS 5 year | 74 (14) | 85 (15)
  EQ-5D VAS 7 year: number analyzed (Participants) | 17 | 20
  EQ-5D VAS 7 year | 78 (15) | 83 (23)
  EQ-5D VAS 10 year: number analyzed (Participants) | 14 | 19
  EQ-5D VAS 10 year | 79 (21) | 83 (15)

5. Secondary Outcome: Investigation of Patient Outcome With Radiographic Analysis
Description: Plain radiographs will be obtained for assessment of fixation of the device.
Time Frame: 3 months, 1, 2, 5, 7 and 10 years
Population: Plain radiographs were used for disease classification. Additional radiographs were not collected for the assessment of device fixation as the RSA analysis was used as an exact measurement of prosthesis components migration and implant fixation.
Arm/Group | Triathlon CR | Triathlon PS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: During entire 10 years follow-up of all patients
Description: All serious adverse events and operative site events occuring in this study were reported.
Arm/Group | Triathlon CR | Triathlon PS
All-Cause Mortality (participants affected / at risk) | 4/28 | 3/30
Serious Adverse Events (participants affected / at risk) | 3/28 | 2/30
Other Adverse Events (participants affected / at risk) | 0/28 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triathlon CR (N=28) | Triathlon PS (N=30)
Total knee replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Contralateral side
Pleomorphic Adenoma of Salivary Glands (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Uterine Cancer
Epileptic fit (Nervous system disorders) | 1 (1) | 0 (0)
Pressure Stroke (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2007-08-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT02522728/Prot_SAP_000.pdf